CLINICAL TRIAL: NCT00431600
Title: The Validity of Retinal Blood Flow Measurements During Hyperoxia in Humans Using Fourier Domain CDOCT
Brief Title: The Validity of Retinal Blood Flow Measurements During Hyperoxia in Humans Using Fourier Domain Color Doppler Optical Coherence Tomography (CDOCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-121103
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: Regional Blood Flow; Color Doppler Optical Coherence Tomography; CDOCT; Retinal Blood Flow; Hyperoxia; Vasoconstriction; Laser Doppler Velocimetry; Retinal Vessel Analyzer
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 12 healthy male subjects
  Interventions: Other: 100% Oxygen

INTERVENTIONS:
Other: 100% Oxygen — 100% Oxygen- breathing over 30 minutes

SUMMARY:
Noninvasive monitoring of blood flow in retinal circulation may elucidate the progression and treatment of ocular disorders, including diabetic retinopathy, age-related macular degeneration and glaucoma.

Laser Doppler velocimetry (LDV), a noninvasive optical method combined with vessel size determination has been used extensively as a valuable research tool to examine blood flow dynamics in the human retina. However, no information on the velocity profile within the vessel is available. Ophthalmic color Doppler optical coherence tomography (CDOCT) provides laser Doppler information in addition to conventional optical coherence tomography, allowing the observation of blood flow dynamics simultaneously to imaging retinal structure.

We have recently demonstrated the feasibility of Fourier domain CDOCT to assess velocity profiles in human retinal vessels in vivo.

In the present study the validity of Fourier domain CDOCT for retinal blood flow measurements will be tested at baseline and during hyperoxia-induced vasoconstriction in humans by comparison with retinal blood flow measurements using a commercially available LDV system and the Zeiss retinal vessel analyzer (RVA)

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 dpt

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Ametropia equal or over 3 dpt

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Retinal blood flow (LDV, RVA) | 15 minutes

SECONDARY OUTCOMES:
Retinal venous diameters (Zeiss retinal vessel analyzer) | 5 minutes
Retinal blood velocity (laser Doppler velocimetry) | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria